CLINICAL TRIAL: NCT03403907
Title: The Effect of Probiotic Supplementation in Drug-resistant Epilepsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: María Gómez Eguílaz (Other Government)
Responsible Party: Sponsor-Investigator, María Gómez Eguílaz, principal investigator, Fundación RiojaSalud
Organization: Fundación RiojaSalud (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: probiotico-epilepsia-001
Record Dates: First submitted 2017-12-21; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy; Epilepsy Intractable
Keywords: epilepsy; microbiota; probiotics
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): Probiotic administration
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Probiotic — twice a day for 4 months (Streptococcus thermophilus, Lactobacillus acidophilus, L.plantarum, L. paracasei, L. delbrueckii subs bulgaricus, Bifidobacterium breve, B.longus y B.infantis. y CD2).

SUMMARY:
This study evaluates the effect of probiotic supplementation in patients with drug-resistant epilepsy. All the patients received the probiotic.

DETAILED DESCRIPTION:
Epilepsy is a neurological disease with a prevalence of 0.6%. Despite the high number of antiepileptic drugs available, 20-30% of patients fail to control their seizures even with a correct treatment, this is known as drug-resistant epilepsy. This type of epilepsy limits severely the quality of life in patients and increases their morbidity and mortality.

There are different therapeutic strategies for the treatment of drug-resistant epilepsy such as the vagus nerve stimulation, which has an effectiveness of approximately 50% reduction of seizures in 50% of patients. Another one is epilepsy surgery, which can achieve up to 70% of crisis control with specifically selected surgery for certain patients. On the other hand, the ketogenic diet has nearly 30% effectiveness, which is defined as a seizure reduction of more than 50%. Despite all these treatments, there is still a group of patients that keeps showing epileptic seizures.

The microbiota is a collective of microorganisms that live in a symbiotic relationship within our organism. Currently, it is known that there is a bidirectional relationship between microbiota-gut-brain. Probiotics are live microorganisms that can benefit the health of the host when administered in adequate doses.

The purpose of the study is to prove the quality of life improvement in drug-resistant patients after the administration of a probiotic for 4 months in order to reduce the number of seizures. Additionally, the parameters of inflammatory cytokines will be evaluated as well as the probiotic medication safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old.
* Diagnosis of drug-resistant epileptic seizures.
* Under stable treatment with antiepileptic drugs for at least 30 days before their inclusion.
* Occurrence of at least one seizure per month.
* Acceptance and informed consent for the inclusion of the patient in the study protocol.

Exclusion Criteria:

* Stable epilepsy.
* Idiopathic generalized epilepsy.
* Epileptic status in the previous 12 months.
* Change in the dose or type of antiepileptic drug within 30 days prior to the start of the study.
* Active consumption of alcohol or substances of abuse.
* Pregnancy and / or mothers during lactation period.
* Patients treated with probiotics from 30 days before the start of the study.
* Chronic gastrointestinal problems (for example irritable bowel).
* Liver or kidney problems.
* Lactose intolerant or celiac.
* Immunosuppressed.
* Patients on chronic antibiotic treatment.
* Impossibility to fill in a questionnaire, by the patient or the person responsible, and to follow the schedule of visits.
* Progressive neurological deterioration (tumors or metastasis of the central nervous system (CNS), Alzheimer's disease, vascular dementias).
* Use of antiepileptic drugs in research.
* Patients with an expectation of life <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of probiotics for controlling epileptic seizures in patients with drug-resistant epilepsy | From visit 2 to visit 3 (administration of probiotics, 4 months)
  effectiveness can be defined as the reduction in number of seizures of at least 50%

SECONDARY OUTCOMES:
Quality of life | From visit 2 to visit 3 (administration of probiotics, 4 months)
  Measured by the questionnaire of quality of life in epilepsy (QOLIE-10) in Spanish language 10-item questionnaire for screening quality-of-life issues for patients with epilepsy, in clinical practice. It evaluates: epilepsy effects, mental health and role function.
  The minimum of scale is 10-maximun: 50 10-19: very well; could hardly be better 20-29: pretty good 30-39: godd and bad parts about equal 40-49: pretty bad 50: very bad; could hardly be worse
Assessing the anti-inflammatory effect of probiotics | From visit 2 to visit 3 (administration of probiotics, 4 months)
  To evaluate inflammatory markers: interleukin-6 (IL-6) and soluble CD14 (sCD14) in blood test.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | From visit 2 to visit 3 (administration of probiotics, 4 months)
  Adverse events monitoring during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: María Gómez Eguílaz, Principal Investigator — Fundación RiojaSalud

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Tojo R, Suarez A, Clemente MG, de los Reyes-Gavilan CG, Margolles A, Gueimonde M, Ruas-Madiedo P. Intestinal microbiota in health and disease: role of bifidobacteria in gut homeostasis. World J Gastroenterol. 2014 Nov 7;20(41):15163-76. doi: 10.3748/wjg.v20.i41.15163. PMID 25386066
- [Derived] Gomez-Eguilaz M, Ramon-Trapero JL, Perez-Martinez L, Blanco JR. The beneficial effect of probiotics as a supplementary treatment in drug-resistant epilepsy: a pilot study. Benef Microbes. 2018 Dec 7;9(6):875-881. doi: 10.3920/BM2018.0018. Epub 2018 Sep 10. PMID 30198325